CLINICAL TRIAL: NCT00782002
Title: Phase 1 Study of Weekly Anti-Vascular Endothelial Growth Factor Receptor 1 (VEGFR-1) Monoclonal Antibody IMC-18F1 in Patients With Advanced Solid Tumors Who No Longer Respond to Standard Therapy or For Whom No Standard Therapy is Available
Brief Title: Safety Study of IMC-18F1,to Treat Advanced Solid Tumors in Subjects That no Longer Respond to Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13941; CP14-0501 (Other: ImClone, LLC); I4Y-IE-JCDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2010-09

CONDITIONS: Advanced Solid Tumors
Keywords: Solid Tumors; VEGF-A; stromal cells; endothelial cells; malignant cells
MeSH Terms: interventions — IMC-18F1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMC-18F1 (Experimental)
  Interventions: Biological: IMC-18F1

INTERVENTIONS:
Biological: IMC-18F1 — Cohorts 1-4 will receive IMC-18F1 intravenously for 4 weekly infusions, followed by a 2-week observation period. Cohort 5 will receive IMC-18F1 intravenously every other week for the first 6 weeks of therapy. Cohort 6 will receive IMC-18F1 every 3 weeks for the first 6 weeks for therapy. The starting dose in Cohort 1 will be 2mg/kg. The maximum dose of IMC-18F1 will not exceed 16mg/kg administered every week, 15mg/kg administered every other week, and 20mg/kg administered every 3 weeks. Dose escalation of 100% (2 x previous dose) if no dose limiting toxicities (DLTs) are observed in the first three patients within a cohort during the initial 6-week therapy period. Dose escalation increment will be reduced to 50% (1.5 x previous dose) following the occurrence of either grade 2 or higher AEs in 2 or more patients that are possibly, probably, or definitely-related to study medication or one DLT during the initial 6-week therapy period. No intrapatient dose escalation is allowed.

SUMMARY:
The purpose of this study is to determine if IMC-18F1 is safe for patients, and also to determine the best dose of IMC-18F1 to give to patients.

DETAILED DESCRIPTION:
The purpose of this study will be to establish the safety profile and the maximum tolerated dose (MTD) of the anti-VEGFR-1 monoclonal antibody IMC-18F1 administered weekly, every other week, or every three weeks in patients with advanced solid tumors who have not responded to standard therapy or for whom no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histopathologically-documented, measurable or non measurable {evaluable}, advanced solid tumors refractory to standard therapy or for which no standard therapy is available (see Section 10.2, Tumor Response, for the definition of measurable and non measurable {evaluable} disease).
2. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2 at study entry.
3. Able to provide written informed consent.
4. Age 18 years or older.
5. A life expectancy of >3 months.
6. Adequate hematologic function, as defined by:

   * an absolute neutrophil count ≥1500/mm3
   * a hemoglobin level ≥ 9gm/dL
   * a platelet count ≥100,000/mm3
7. Adequate hepatic function, as defined by:

   * a total bilirubin level ≤1.5 x the ULN
   * aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤2.5 x the ULN or ≤5 x the ULN if known liver metastases
8. Adequate renal function, as defined by a serum creatinine level ≤1.5 x the ULN.
9. Use of effective contraception (per the institutional standard), if procreative potential exists.
10. Adequate recovery from recent surgery, chemotherapy, and radiation therapy. At least 28 days must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, or prior radiation therapy (palliative radiation therapy is allowed).
11. Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center.

Exclusion Criteria:

1. Patients who have had chemotherapy or therapeutic radiotherapy within 28 days prior to entering the study or patients with ongoing side effects ≥ grade 2 due to agents administered more than 28 days earlier.
2. Uncontrolled intercurrent illness including, but not limited to:

   * ongoing or active infection requiring parenteral antibiotics
   * symptomatic congestive heart failure (class III or IV of the New York Heart Association classification for heart disease)
   * left ventricular ejection fraction (LVEF) of <50%. If a baseline MUGA shows a <50% ejection fraction, then a confirmatory ultrasound should be performed. If it is <50%, the patient is excluded from the study
   * unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
   * uncontrolled hypertension (systolic blood pressure >150 mm Hg, diastolic blood pressure >100 mm Hg, found on two consecutive measurements separated by a 1-week period despite adequate medical support)
   * clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment [Common Terminology Criteria for Adverse Events {CTCAE}, Version 3.0, grade 3] or asymptomatic sustained ventricular tachycardia)
   * uncontrolled diabetes
   * psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements
3. Patients with progressive or symptomatic brain or leptomeningeal metastases. (Patients with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and not taking steroids; anti-seizure medications are allowed).
4. A serious or nonhealing active wound, ulcer, or bone fracture.
5. Known human immunodeficiency virus positivity.
6. A major surgical procedure, an open biopsy, or a significant traumatic injury within 28 days prior to treatment.
7. Current or recent use (within 28 days) of a thrombolytic agent.
8. Current use of full-dose warfarin (an exception is low-dose warfarin to maintain patency of pre-existing, permanent, indwelling intravenous (i.v.) catheters; for patients receiving warfarin, the international normalized ratio [INR] should be <1.5), heparin or fractionated heparin are excluded.
9. Chronic daily treatment with aspirin (>325 mg/day), nonsteroidal antiinflammatory or other medications known to inhibit platelet function (cyclooxygenase-2 [COX-2] inhibitors are permitted).
10. A history or clinical evidence of a deep venous or arterial thrombosis (including pulmonary embolism) within 6 months prior to study entry.
11. Proteinuria ≥2+ by routine urinalysis or dipstick and subsequent documentation by 24-hour urine collection of >1 g protein. Patients with genitourinary malignancies and/or those with a requirement for urinary catheters or stents will be excluded if the 24-hour urine protein is ≥2 g.
12. Pregnant (confirmed by serum beta human chorionic gonadotropin [βHCG]) or breast feeding.
13. Positive for anti-IMC-18F1 antibodies.
14. Treatment with monoclonal antibodies within 6 weeks of study entry.
15. A history of allergic reactions to monoclonal antibodies or other therapeutic proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-07; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 6 weeks

SECONDARY OUTCOMES:
Pharmacokinetics | 6 weeks
Antitumor Activity of IMC-18F1 Monotherapy | 6 Weeks
Pharmacodynamics | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - ImClone Investigational Site, Detroit, Michigan
  - ImClone Investigational Site, Cleveland, Ohio

REFERENCES:
- [Derived] LoRusso PM, Krishnamurthi S, Youssoufian H, Hall N, Fox F, Dontabhaktuni A, Grebennik D, Remick S. Icrucumab, a fully human monoclonal antibody against the vascular endothelial growth factor receptor-1, in the treatment of patients with advanced solid malignancies: a Phase 1 study. Invest New Drugs. 2014 Apr;32(2):303-11. doi: 10.1007/s10637-013-9998-8. Epub 2013 Aug 1. PMID 23903897